CLINICAL TRIAL: NCT01547455
Title: Anti-inflammatory and Renoprotective Effect of Pretreatment Loading Dose Atorvastatin in CABG
Brief Title: Safety and Efficiency Study of Loading Dose Atorvastatin in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Shan Zhou, Principal Investigator, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-1002-007
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Acute Kidney Injury
Keywords: Statin; kidney function; antiinflammatory effect
MeSH Terms: conditions — Acute Kidney Injury | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): participants take 80mg Atorvastatin orally 12h before surgery with another 40mg 2h before surgery
  Interventions: Drug: Atorvastatin(Lipitor)
- Control (Placebo Comparator): Participants randomized to Control arm take 80mg placebo 12h before surgery with another 40mg 2h before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin(Lipitor) — participants take 80mg Atorvastatin orally 12h before surgery with another 40mg 2h before surgery
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — Participants randomized to Control arm take 80mg placebo 12h before surgery with another 40mg 2h before surgery
  Arms: Control

SUMMARY:
Statins were reported to have pleiotropic effects including antiinflammatory, anti-oxidative stress effects and stabilise plaque in some conditions. Some researches indicate loading dose statin can reduce contrast induced nephropathy, and the levels of inflammatory markers were significantly decreased. The investigators hypothesis loading dose atorvastatin may attenuate inflammatory response during cardiopulmonary bypass (CPB) and therefore reduce postoperative acute kidney injury in cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury occurs up to 30% in cardiac surgery which influenced patients' mid-term and long-term outcomes. Furthermore, evidence shows patients who initiate renal placement therapy in hospital have higher mortality and morbility. The pathologies of Cardiac surgery-associated acute kidney injury (CSA-AKI) is not clear yet ,many researches find cardiopulmonary bypass is an independent risk factor in developing AKI, and inflammatory bursts during cardiopulmonary bypass (CPB) may play an important role in CSA-AKI.

Statins are reported to have anti-inflammatory reaction in many researches. In Some multicenter RCTS, Statins are reported to reduce myocardial infarction,atrial fibrillation and have renoprotective effects due to pleiotropic effects in percutaneous coronary intervention. While in the cardiac surgery settings, the renoprotective effect of statin is still controversial. The investigators believe the differences between surgery and PCI may contribute to the discrepancy. The investigators plan to test the renoprotective effect of atorvastatin in a randomized,double-blind control manner and try to explore the mechanism of this protective effect.

The investigators hypothesise loading dose atorvastatin pretreatment in elective coronary artery bypass grafting surgery may attenuate inflammatory response in CPB and therefore reduce postoperative AKI or help recovery from AKI.

The investigators randomize patients into two arms, the Atorvastatin group takes Atorvastatin 80mg 12h before surgery with another 40mg 2h before operation, the control arm takes placebo in the same regime. The investigators plan to compare the inflammatory cytokines at different time points and the incidence of AKI between the two groups. The investigators hope Atorvastatin group can decrease AKI incidence and has a lower level of inflammatory cytokines, what's more, the two have a good correlation in the time frame.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* elective coronary artery bypass surgery in CPB

Exclusion Criteria:

* emergent surgery
* re-operation
* acute kidney dysfunction
* chronic kidney disease
* GFR < 60ml/min
* liver dysfunction
* existing myopathy
* LEVF < 40%
* statin allergic or contradictive
* pregnancy
* breast feed period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | 72 hours after surgery
  Proportion developing AKI using AKIN criteria(stage 1,stage 2, stage3).we plan to measure serum creatinine in baseline, ICU admission,postoperative 6h、Day 1、Day 2 and Day 3.If multiple SCr was measured in one day ,then the highest value will be recorded.Also, we measure creatinine clearance via Cock-croft-Gault formula.

SECONDARY OUTCOMES:
Change of inflammatory biomarkers | 48h after surgery
  we plan to measure IL-6,IL-10,TNF-α and hsCRP at 6 time points: before surgery、after chest closure、postOp.6h、12h、24h and 48h.Compare levels of cytokines between the two arms
Requirement of renal replacement therapy | participants will be followed for the duration of hospital stay , an expected average of 2 weeks
  proportion need renal replacement therapy in hospital
liver function | participants will be followed for the duration of hospital stay , an expected average of 2 weeks
  liver dysfunction defined as transaminase>3UNL normal level
death | 30 days after discharge from hospital
MACCE events | 30 days after discharge from hospital
length of stay in intensive care unit | From admission to discharge from ICU
  An average of 2 days
length of stay in hospital after surgery | From surgery to discharge from hospital, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Weipeng Wang, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Cardiovascular Institute&Fuwai Hospital, Beijing, Beijing Municipality, China